CLINICAL TRIAL: NCT04963270
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study To Evaluate Efficacy, Safety, Pharmacokinetics, And Pharmacodynamics Of Satralizumab In Patients With Generalized Myasthenia Gravis
Brief Title: A Study To Evaluate Efficacy, Safety, Pharmacokinetics, And Pharmacodynamics Of Satralizumab In Patients With Generalized Myasthenia Gravis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to halt development of satralizumab in generalized myasthenia gravis and discontinued further dosing with the study drug (while the OLE period was ongoing) upon reviewing the primary results (DB period).
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN42636
Record Dates: First submitted 2021-07-07; First posted 2021-07-15 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — satralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Satralizumab (Experimental): Participants will receive Satralizumab at Weeks 0, 2, 4, and Q4W thereafter. Adolescent patients who first enter the study in the OLE period will receive satralizumab SC loading doses at Week 0, 2, and 4 in the OLE, followed by maintenance doses Q4W thereafter and will remain on stable background therapy until Week 24 of the OLE.
  Interventions: Drug: Satralizumab
- Placebo (Placebo Comparator): Participants will receive placebo at Weeks 0, 2, 4, and Q4W thereafter
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Satralizumab — Satralizumab will be administered as a subcutaneous injection
  Arms: Satralizumab
Other: Placebo — Satralizumab placebo will be administered as a subcutaneous injection
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of satralizumab compared with placebo in participants with generalized myasthenia gravis (gMG).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* For adolescent patients: Informed Consent Form for study participation signed by the parents or a legal guardian, and patient assent obtained, as per local requirements
* Ability to comply with the study protocol procedures
* Confirmed diagnosis of gMG (anti-AChR, anti-MuSK or anti-LRP4 present at screening)
* A total MG-ADL score of ≥ 5 points at screening with more than 50% of this score attributed to non-ocular items
* MGFA severity Class II-IV
* Ongoing gMG treatment at a stable dose
* For female patients of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate contraception during the treatment period and for at least 3 months after the final dose of satralizumab.

Exclusion Criteria:

* History of thymectomy within 12 months prior to screening
* Ocular MG (MGFA Class I) and myasthenic crisis (MGFA Class V) within the last 3 months prior to screening
* Known disease other than gMG that would interfere with the course and conduct of the study
* Positive screening tests for hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Evidence of latent or active tuberculosis (excluding patients receiving chemoprophylaxis for latent tuberculosis infection)
* Receipt of live or live attenuated vaccine within 6 weeks prior to baseline
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the last dose

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (76):
- United States (6):
  - Keck School of Medicine of USC, Los Angeles, California
  - University of California Irvine - Manchester Pavilion, Orange, California
  - SC3 Research Group, Inc, Pasadena, California
  - Medical Faculty Associates Inc., Washington D.C., District of Columbia
  - University of Chicago Hospital, Chicago, Illinois
  - Prairie Education and Research, O'Fallon, Illinois
- Argentina (5):
  - Hospital Italiano, CABA
  - Hospital Ramos Mejía, CABA
  - Hospital Britanico, Ciudad Autonoma Bs As
  - Fundación Scherbovsky, Mendoza
  - INECO Neurociencias Orono, Rosario
- Concord Repatriation General Hospital, Concord, New South Wales, Australia
- Brazil (4):
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Hospital Sao Paulo, São Paulo, São Paulo
- MUCH - Montreal Neurological Institute & Hospital, Montreal, Quebec, Canada
- China (12):
  - Beijing Tongren Hospital, Beijing
  - Beijing Tiantan Hospital,Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital - Sichuan University, Chengdu
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Sir Run Run Shaw Hospital, Hangzhou
  - The First Affiliated Hospital Of Shandong First Medical University, Jinan
  - Huashan Hospital, Fudan University, Shanghai
  - Children's Hospital of Fudan University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tangdu Hospital, Xi'an
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, København Ø
- France (5):
  - CHU Bordeaux, Bordeaux
  - APHP Raymond Poincare, Garches
  - Hopital Timone Adultes, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU Nice - Hôpital Pasteur 2, Nice
- Germany (3):
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Universitätsklinikum Essen (AöR), Essen
  - Universitätsklinikum Münster, Münster
- Italy (4):
  - Azienda Ospedaliera A. Cardarelli, Napoli, Campania
  - Fond. Istituto Neurologico C.Besta, Milan, Lombardy
  - A.R.N.A.S. Civico Di Cristina Benfratelli, Palermo, Sicily
  - Ospedale Cà Foncello, Treviso, Veneto
- Japan (12):
  - Juntendo University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba-shi, Chiba
  - General Hanamaki Hospital, Hanamaki, Iwate
  - Sapporo Medical University Hospital, Hokkaido
  - NHO Hokkaido Medical Center, Hokkaido
  - St. Marianna University Hospital, Kanagawa
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Kindai University Hospital, Osaka
  - Seirei Hamamatsu General Hospital, Shizuoka
  - Osaka University Hospital, Suita
  - Tokyo Medical And Dental University, Medical Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Poland (4):
  - Klinika Neurologii Doros?ych, Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Zespol Poradni Specjalistycznych - Poradnia Neurologiczna, Krakow
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii K, Krakow
  - Indywidualna Praktyka Lekarska Prof. Dr Hab. N. Med. Konrad Rejdak., Lublin
- Russia (2):
  - Krasnoyarsk State Medical Academy, Krasnoyarsk, Krasnoyarsk Krai
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
- South Korea (5):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (4):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario la Fe, Valencia
- Taiwan (2):
  - Taipei Veterans General Hospital-Neurology, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
- Turkey (Türkiye) (4):
  - Hacettepe University Medical Faculty, Ankara
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Hospital, Kocaeli
  - Ondokuz Mayis Univ. Med. Fac., Samsun

REFERENCES:
- [Derived] Habib AA, Zhao C, Aban I, Franca MC Jr, Jose JG, Zu Horste GM, Klimiec-Moskal E, Pulley MT, Tavolini D, Krumova P, Lennon-Chrimes S, Smith J, Thanei GA, Blondeau K, Vodopivec I, Wolfe GI, Murai H. Safety and efficacy of satralizumab in patients with generalised myasthenia gravis (LUMINESCE): a randomised, double-blind, multicentre, placebo-controlled phase 3 trial. Lancet Neurol. 2025 Feb;24(2):117-127. doi: 10.1016/S1474-4422(24)00514-3. PMID 39862880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 188 participants with generalized myasthenia gravis (gMG) took part in the study across 76 investigational sites in 17 countries. Of the 188, 2 adolescent participants were randomized after the last adult participant was enrolled in the study and therefore were not part of efficacy analysis.
Pre-assignment Details: The study consists of 2 periods: Double-blind (DB) period where participants were randomized in a 1:1 ratio to receive either satralizumab or matching placebo and an open-label extension (OLE) period where all participants who completed the DB period received satralizumab. Participants were on a stable dose of background therapy (for gMG) throughout the DB period and until Week 12 of the OLE period.
Groups:
- Placebo: Participants received satralizumab matched placebo, subcutaneously (SC), at Weeks 0, 2, 4, and every 4 weeks (Q4W) thereafter until the end of the DB period.
- Satralizumab: Participants received satralizumab 120 (milligrams) mg or 180 mg, based on body weight, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
- Placebo (DB) to Satralizumab (OLE): After completion of the DB period, participants entered the OLE period where they received satralizumab, 120 mg or 180 mg, based on body weight, SC at Weeks 0, 2, and 4 (loading doses), and Q4W thereafter (maintenance doses) during the OLE period.
- Satralizumab (DB) to Satralizumab (OLE): After completion of the DB period, participants entered the OLE period and continued receiving satralizumab 120 mg or 180 mg, based on body weight, SC until the end of the OLE period. Participants received a placebo injection on Week 2 of OLE to maintain blinding to DB treatment assignment.
Period: Double-Blind Period (24 Weeks)
Arm/Group | Placebo | Satralizumab | Placebo (DB) to Satralizumab (OLE) | Satralizumab (DB) to Satralizumab (OLE)
Started | 92 | 96 | 0 | 0
Completed | 88 | 92 | 0 | 0
Not Completed | 4 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 2 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 1 | 0 | 0
Period: Open Label Extension Period (92 Weeks)
Arm/Group | Placebo | Satralizumab | Placebo (DB) to Satralizumab (OLE) | Satralizumab (DB) to Satralizumab (OLE)
Started | 0 | 0 | 88 | 92
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 88 | 92
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 6
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 82 | 81
Not completed — Reason Not Specified | 0 | 0 | 0 | 1
Not completed — Reason Unknown | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Overall Population (OP) included all randomized participants who were either acetylcholine receptor antibody seropositive (AChR+) or acetylcholine receptor antibody seronegative (AChR-).
Groups:
- Placebo: Participants received satralizumab matched placebo, SC, at Weeks 0, 2, 4, and Q4W thereafter until the end of the DB period.
- Satralizumab: Participants received satralizumab 120 mg or 180 mg, based on body weight, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Satralizumab | Total
Number analyzed (Participants) | 92 | 96 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (16.3) | 47.0 (14.4) | 46.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 63 | 119
  Male | 36 | 33 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 24 | 54
  Not Hispanic or Latino | 54 | 70 | 124
  Unknown or Not Reported | 8 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 27 | 32 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 56 | 59 | 115
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Mean Change From Baseline in Total Myasthenia Gravis Activities of Daily Living (MG-ADL) Score in the AChR+ Population
Description: The MG-ADL scale was used to assess the degree of gMG symptoms (six items: diplopia, ptosis, difficulties with chewing, swallowing, talking, and respiratory problems) and functional limitations in carrying out activities of daily living (two items: ability to brush teeth or comb hair and impairment in the ability to arise from a chair) that are present and clinically relevant in gMG participants. Each of the eight items was ranked on a 0-3 scale, with 3 representing the most severe symptoms or impaired performance and 0 representing no symptoms or impaired performance. The total MG-ADL score was calculated as the sum of each item score, with a maximum score ranging from 0 (least severe symptoms/impairment) to 24 (most severe symptoms/impairment). Higher scores indicate greater disease severity.
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
score on a scale | -2.57 (0.35) | -3.59 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0196, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -1.02, 95% CI 2-sided [-1.88 to -0.16], Standard Deviation 0.44

2. Secondary Outcome: DB Period: Mean Change From Baseline in Total MG-ADL Score in the Overall Population (OP) at Week 24
Description: as for outcome 1
Time Frame: At Week 24
Population: Modified intent-to-treat (mIIT) population included all participants that were part of the ITT and had a baseline and at least one post-baseline MG-ADL assessment during the DB period. This excludes adolescents who joined the study after the last adult participant was randomized.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
score on a scale | -2.52 (0.32) | -3.54 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0123, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -1.02, 95% CI 2-sided [-1.82 to -0.22], Standard Error of Mean 0.41

3. Secondary Outcome: DB Period: Percentage of Participants With a ≥ 2-point Reduction From Baseline in Total MG-ADL Score in AChR+ Population at Week 24
Description: The MG-ADL scale was used to assess the degree of gMG symptoms (six items: diplopia, ptosis, difficulties with chewing, swallowing, talking, and respiratory problems) and functional limitations in carrying out activities of daily living (two items: ability to brush teeth or comb hair and impairment in the ability to arise from a chair) that are present and clinically relevant in gMG participants. Each of the eight items was ranked on a 0-3 scale, with 3 representing the most severe symptoms or impaired performance and 0 representing no symptoms or impaired performance. The total MG-ADL score was calculated as the sum of each item score, with a maximum score ranging from 0 (least severe symptoms/impairment) to 24 (most severe symptoms/impairment). Higher scores indicate greater disease severity. Participants who received rescue therapy were considered non-responders.
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
percentage of participants | 58.8 [47.9 to 69.6] | 70.9 [61.2 to 80.6]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Stratified Analysis; Test type: Superiority; p = 0.088, Cochran-Mantel-Haenszel; Difference in Response Rate = -12.7, 95% CI 2-sided [-27.3 to 1.9]

4. Secondary Outcome: DB Period: Percentage of Participants With a ≥ 2-point Reduction From Baseline in Total MG-ADL Score in OP at Week 24
Description: as for outcome 3
Time Frame: At Week 24
Population: mIIT population included all participants that were part of the ITT and had a baseline and at least one post-baseline MG-ADL assessment during the DB period. This excludes adolescents who joined the study after the last adult participant was randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
percentage of participants | 60.7 [50.4 to 70.9] | 69.8 [60.5 to 79]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Stratified Analysis; Test type: Superiority; p = 0.137, Cochran-Mantel-Haenszel; Difference in Response Rate = -10.5, 95% CI 2-sided [-24.2 to 3.3]

5. Secondary Outcome: DB Period: Mean Change From Baseline in Quantitative Myasthenia Gravis (QMG) Score in AChR+ Population at Week 24
Description: The QMG is a 13-item direct physician assessment scoring system that quantifies disease severity based on impairments of body functions and structures. The 13-items are: ptosis, diplopia, orbicularis oculi weakness, swallowing, speech disruption, percent forced vital capacity, arm and leg endurance (four items), grip strength (two items), and neck flexion strength. Each of the 13 item was quantitatively assessed and scored on a scale from 0=None to 3=Severe, providing a total QMG score (sum of each item score) ranging from 0 to 39 where higher scores indicate greater disease severity.
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
score on a scale | -1.78 (0.46) | -3.41 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0062, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -1.63, 95% CI 2-sided [-2.80 to -0.46], Standard Error of Mean 0.60

6. Secondary Outcome: DB Period: Mean Change From Baseline in QMG Score in OP at Week 24
Description: as for outcome 5
Time Frame: At Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
score on a scale | -1.74 (0.43) | -3.42 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0034, ANCOVA and Conditional Mean Imputation; Difference in adjusted Mean = -1.68, 95% CI 2-sided [-2.80 to -0.56], Standard Error of Mean 0.57

7. Secondary Outcome: DB Period: Mean Change From Baseline in Myasthenia Gravis Quality of Life 15 Scale (Revised) (MG-QOL 15r) Total Score in AChR+ Population at Week 24
Description: The MG-QOL-15r is a disease-specific health-related QoL measure that consists of 15 items: mobility (9 items), symptoms (3 items), and contentment and emotional well-being (3 items). Items were scored on a scale from 0=Not at all to 2=Very much with the total score ranging from 0 to 30 and higher scores indicate worse health-related quality of life (HRQoL).
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
score on a scale | -4.69 (0.71) | -6.20 (0.69)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.1094, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -1.51, 95% CI 2-sided [-3.36 to 0.34], Standard Error of Mean 0.94

8. Secondary Outcome: DB Period: Mean Change From Baseline in MG-QOL 15r Total Score in OP at Week 24
Description: The MG-QOL-15r is a disease-specific health-related QoL measure that consists of 15 items: mobility (9 items), symptoms (3 items), and contentment and emotional well-being (3 items). Items are scored on a scale from 0=Not at all to 2=Very much, with the total score ranging from 0 to 30 and higher scores indicate worse HRQoL.
Time Frame: At Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
score on a scale | -4.73 (0.65) | -6.13 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0999, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -1.39, 95% CI 2-sided [-3.05 to 0.27], Standard Error of Mean 0.85

9. Secondary Outcome: DB Period: Mean Change From Baseline in Quality of Life in Neurological Disorders (Neuro-QoL) Fatigue Subscale Total Score in AChR+ Population at Week 24
Description: The Neuro-QoL is a validated tool designed to evaluate the HRQoL in participants with chronic neurological disease. The Fatigue Subscale is implemented as an eight-item, stand-alone short form that assesses the multi-dimensional aspects of fatigue ranging from general tiredness to debilitating exhaustion that Impacts activities of daily living. Each item was assessed using a 5-level Likert scale ranging between 1=never to 5=always. Raw scores range from 8 to 40, higher values indicate greater fatigue.
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
score on a scale | -3.29 (0.90) | -5.50 (0.75)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0456, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -2.20, 95% CI 2-sided [-4.36 to -0.04], Standard Error of Mean 1.10

10. Secondary Outcome: DB Period: Mean Change From Baseline in Neuro-QoL Fatigue Subscale Total Score in OP at Week 24
Description: as for outcome 9
Time Frame: At Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
score on a scale | -3.45 (0.83) | -5.56 (0.69)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0382, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -2.11, 95% CI 2-sided [-4.10 to -0.11], Standard Error of Mean 1.02

11. Secondary Outcome: DB Period: Percentage of Participants With a ≥ 3-point Reduction From Baseline in QMG Score in AChR+ Population at Week 24
Description: as for outcome 5
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
percentage of participants | 28.7 [18.7 to 38.8] | 47.7 [37 to 58.3]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority — Stratified Analysis; p = 0.013, Cochran-Mantel-Haenszel; Difference in Response Rate = -18.7, 95% CI 2-sided [-33.5 to -3.9]

12. Secondary Outcome: DB Period: Percentage of Participants With a ≥ 3-point Reduction From Baseline in QMG Score in OP at Week 24
Description: as for outcome 5
Time Frame: At Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
percentage of participants | 28.1 [18.7 to 37.5] | 50.0 [39.9 to 60.1]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority — Stratified Analysis; p = 0.002, Cochran-Mantel-Haenszel; Difference in Response Rate = -22, 95% CI 2-sided [-36.2 to -7.9]

13. Secondary Outcome: DB Period: Mean Change From Baseline in Total Myasthenia Gravis Composite (MGC) Score in AChR+ Population at Week 24
Description: The MGC is a composite measure consisting of items drawn from the MG-ADL (chewing, swallowing, speech, and breathing), QMG (diplopia and ptosis), and Manual Muscle Test (hip flexion strength, neck, facial, and shoulder abduction) in an effort to include both clinician- and participant-reported elements in a single measure. Each of the ten items contribute to a total score ranging from 0 to 50, with higher values indicating greater disease severity.
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
score on a scale | -4.14 (0.62) | -7.13 (0.58)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0002, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -2.99, 95% CI 2-sided [-4.57 to -1.41], Standard Error of Mean 0.81

14. Secondary Outcome: DB Period: Mean Change From Baseline in Total MGC Score in OP at Week 24
Description: as for outcome 13
Time Frame: At Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
score on a scale | -4.18 (0.57) | -7.18 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p < 0.0001, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = -3.00, 95% CI 2-sided [-4.47 to -1.53], Standard Error of Mean 0.75

15. Secondary Outcome: DB Period: Percentage of Participants With a ≥ 3-point Reduction From Baseline in Total MGC Score in AChR+ Population at Week 24
Description: as for outcome 13
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
percentage of participants | 55.0 [44 to 66] | 75.6 [66.4 to 84.7]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Difference in Response Rate = -21, 95% CI 2-sided [-35.4 to -6.6]

16. Secondary Outcome: DB Period: Percentage of Participants With a ≥ 3-point Reduction From Baseline in Total MGC Score in OP at Week 24
Description: as for outcome 13
Time Frame: At Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
percentage of participants | 57.3 [46.9 to 67.7] | 76.0 [67.4 to 84.6]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority — Stratified Analysis; p = 0.005, Cochran-Mantel-Haenszel; Difference in Response Rate = -19.4, 95% CI 2-sided [-32.8 to -5.9]

17. Secondary Outcome: DB Period: Percentage of Participants Who Achieved Minimal Symptom Expression (Total MG-ADL Score of 0 or 1) in AChR+ Population at Week 24
Description: as for outcome 1
Time Frame: At Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
percentage of participants | 12.5 [-4.8 to 29.8] | 14.0 [6.6 to 21.3]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.847, Cochran-Mantel-Haenszel; Difference in Response Rate = -1.7, 95% CI 2-sided [-19.4 to 15.9]

18. Secondary Outcome: DB Period: Percentage of Participants Who Achieved Minimal Symptom Expression (Total MG-ADL Score of 0 or 1) in OP at Week 24
Description: as for outcome 1
Time Frame: At Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
percentage of participants | 12.4 [4.2 to 20.5] | 15.6 [8.3 to 22.9]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority — Stratified Analysis; p = 0.441, Cochran-Mantel-Haenszel; Difference in Response Rate = -4.3, 95% CI 2-sided [-15.4 to 6.7]

19. Secondary Outcome: DB Period: Percentage of Participants With at Least One gMG-Related Exacerbation Between Baseline and Week 24 in AChR+ Population
Description: gMG-related exacerbation was defined as one of the following: MG crisis; Substantial symptomatic worsening that requires immediate therapy; or health in jeopardy if rescue therapy is not given.
Time Frame: Baseline up to Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
percentage of participants | 17.5 [9.1 to 25.9] | 9.3 [3.1 to 15.5]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.115, Cochran-Mantel-Haenszel; Difference in Response Rate = 8.5, 95% CI 2-sided [-2.1 to 19]

20. Secondary Outcome: DB Period: Percentage of Participants With at Least One gMG-Related Exacerbation Between Baseline and Week 24 in OP
Description: as for outcome 19
Time Frame: Baseline up to Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
percentage of participants | 16.9 [9 to 24.7] | 8.3 [2.8 to 13.9]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority — Stratified Analysis; p = 0.077, Cochran-Mantel-Haenszel; Difference in Response Rate = 8.8, 95% CI 2-sided [-1 to 18.6]

21. Secondary Outcome: DB Period: Percentage of Participants in AChR+ Population Receiving Rescue Therapy Between Baseline and Week 24
Description: The percentage of participants receiving rescue therapy during DBP analyzed the variable that encodes whether a participant received rescue therapy during DBP or not. If a participant stopped the study drug but received rescue therapy during the safety follow-up and this occurred within 24 weeks of baseline then this was counted as having received rescue therapy.
Time Frame: Baseline up to Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
percentage of participants | 13.8 [5.58 to 21.92] | 7.0 [1.01 to 12.94]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.1314, Cochran-Mantel-Haenszel; Risk Difference = -6.77, 95% CI 2-sided [-17.25 to 3.70]

22. Secondary Outcome: DB Period: Percentage of Participants in OP Receiving Rescue Therapy Between Baseline and Week 24
Description: as for outcome 21
Time Frame: Baseline up to Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
percentage of participants | 12.4 [4.96 to 19.76] | 7 [1.57 to 13.01]
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority — Stratified Analysis; p = 0.2264, Cochran-Mantel-Haenszel; Risk Difference = -5.07, 95% CI 2-sided [-14.74 to 4.61]

23. Secondary Outcome: DB Period: Duration of Meaningful Improvement, Defined as ≥ 2-Point Reduction From Baseline in Total MG-ADL Score in AChR+ Population
Description: The duration was the difference in weeks between the two visits defining the start and end (or Week 24) of reduction from baseline. The MG-ADL scale was used to assess the degree of gMG symptoms (six items: diplopia, ptosis, difficulties with chewing, swallowing, talking, and respiratory problems) and functional limitations in carrying out activities of daily living (two items: ability to brush teeth or comb hair and impairment in the ability to arise from a chair) that are present and clinically relevant in gMG participants. Each of the eight items was ranked on a 0-3 scale, with 3 representing the most severe symptoms or impaired performance and 0 representing no symptoms or impaired performance. The total MG-ADL score was calculated as the sum of each item score, with a maximum score ranging from 0 (least severe symptoms/impairment) to 24 (most severe symptoms/impairment). Higher scores indicate greater disease severity.
Time Frame: Baseline, Week 24
Population: AChR+ population included all participants in the study who were AChR+.
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 80 | 86
weeks | 7.46 (1.00) | 10.90 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority; p = 0.0179, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = 3.44, 95% CI 2-sided [0.59 to 6.29], Standard Error of Mean 1.45

24. Secondary Outcome: DB Period: Duration of Meaningful Improvement, Defined as ≥ 2-Point Reduction From Baseline in Total MG-ADL Score in OP
Description: as for outcome 23
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Placebo | Satralizumab
Number analyzed (Participants) | 89 | 96
weeks | 7.29 (0.95) | 11.02 (0.98)
Statistical Analysis 1: Comparison: Placebo vs Satralizumab; Test type: Superiority — Stratified Analysis; p = 0.0066, ANCOVA and Conditional Mean Imputation; Difference in Adjusted Mean = 3.73, 95% CI 2-sided [1.04 to 6.42], Standard Error of Mean 1.37

25. Secondary Outcome: DB Period: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptoms, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Day 1 up to approximately 24 weeks
Population: Safety-evaluable (SE) population included all enrolled participants who received at least one dose of study drug, with participants grouped according to treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Satralizumab 120 mg: Participants received satralizumab 120 mg, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
- Satralizumab 180mg: Participants received satralizumab 180 mg, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
Arm/Group | Placebo | Satralizumab 120 mg | Satralizumab 180mg
Number analyzed (Participants) | 92 | 87 | 9
Participants | 67 | 78 | 8

26. Secondary Outcome: DB Period: Serum Levels of Interleukin-6 (IL-6)
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20 and 24
Population: SE Population included all enrolled participants who received at least one dose of study drug, with participants grouped according to treatment received. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters (ng/mL)
Groups:
- Placebo Matched to 120 mg Satralizumab; Placebo Matched to 180 mg Satralizumab: Participants received placebo matched to satralizumab, SC, at Weeks 0, 2, 4, and Q4W thereafter until the end of the DB period.
- Satralizumab 120 mg: Participants received satralizumab 120 mg, based on body weight, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
- Satralizumab 180 mg: Participants received satralizumab 180 mg, based on body weight, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
Arm/Group | Placebo Matched to 120 mg Satralizumab | Satralizumab 120 mg | Placebo Matched to 180 mg Satralizumab | Satralizumab 180 mg
Number analyzed (Participants) | 75 | 87 | 16 | 9
nanograms/milliliters (ng/mL)
  Baseline | 1.97 (70.7) | 2.19 (79.3) | 3.65 (124.3) | 4.87 (87.7)
  Week 2: number analyzed (Participants) | 71 | 83 | 16 | 8
  Week 2 | 2.30 (90.8) | 17.45 (100.6) | 3.08 (118.5) | 35.23 (91.8)
  Week 4: number analyzed (Participants) | 73 | 86 | 16 | 9
  Week 4 | 2.10 (81.0) | 20.31 (119.7) | 2.66 (63.3) | 46.49 (87.1)
  Week 8: number analyzed (Participants) | 75 | 84 | 16 | 9
  Week 8 | 2.37 (92.3) | 19.40 (100.8) | 2.46 (84.5) | 38.59 (37.9)
  Week 12: number analyzed (Participants) | 69 | 83 | 16 | 8
  Week 12 | 2.11 (78.3) | 16.59 (93.0) | 3.90 (81.4) | 41.72 (45.5)
  Week 16: number analyzed (Participants) | 67 | 80 | 13 | 9
  Week 16 | 2.17 (91.0) | 18.02 (100.2) | 2.65 (71.8) | 30.13 (67.1)
  Week 20: number analyzed (Participants) | 72 | 80 | 16 | 9
  Week 20 | 2.24 (93.4) | 15.50 (112.7) | 2.96 (98.7) | 26.10 (220.1)
  Week 24: number analyzed (Participants) | 71 | 81 | 16 | 9
  Week 24 | 2.18 (99.5) | 15.75 (95.7) | 2.26 (77.1) | 29.57 (161.2)

27. Secondary Outcome: DB Period: Serum Levels of Soluble Interleukin-6 Receptors (sIL-6R)
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20 and 24
Population: SE Population included all enrolled participants who received at least one dose of study drug, with participants grouped according to treatment received. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo Matched to 120 mg Satralizumab | Satralizumab 120 mg | Placebo Matched to 180 mg Satralizumab | Satralizumab 180 mg
Number analyzed (Participants) | 76 | 87 | 16 | 9
ng/mL
  Baseline | 36.39 (27.3) | 35.95 (24.8) | 34.52 (27.9) | 41.90 (24.4)
  Week 2: number analyzed (Participants) | 72 | 85 | 16 | 8
  Week 2 | 36.08 (25.8) | 461.84 (18.1) | 35.51 (24.0) | 441.03 (32.9)
  Week 4: number analyzed (Participants) | 73 | 87 | 16 | 9
  Week 4 | 34.88 (26.0) | 608.26 (18.1) | 35.65 (23.3) | 558.11 (27.3)
  Week 8: number analyzed (Participants) | 75 | 87 | 16 | 9
  Week 8 | 35.26 (27.9) | 659.47 (19.4) | 33.04 (28.1) | 653.33 (23.6)
  Week 12: number analyzed (Participants) | 70 | 84 | 16 | 8
  Week 12 | 36.54 (26.9) | 643.91 (26.3) | 33.45 (26.2) | 646.65 (25.2)
  Week 16: number analyzed (Participants) | 68 | 81 | 14 | 9
  Week 16 | 35.58 (25.1) | 646.92 (25.9) | 35.80 (29.6) | 600.54 (40.2)
  Week 20: number analyzed (Participants) | 73 | 82 | 16 | 9
  Week 20 | 34.58 (24.6) | 637.30 (23.9) | 33.30 (24.8) | 430.87 (124.1)
  Week 24: number analyzed (Participants) | 71 | 83 | 16 | 9
  Week 24 | 37.46 (58.7) | 634.58 (25.8) | 34.12 (24.1) | 374.27 (158.9)

28. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) to Satralizumab
Description: The percentage of ADA-positive participants after drug administration were determined for participants exposed to satralizumab. For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the baseline titer result. Participants were considered to be ADA-negative if they were ADA-negative or had missing data at baseline and all post-baseline samples were negative, or if they were ADA positive at baseline but did not have any post-baseline samples with a titer that is at least 4-fold (0.60 titer unit) greater than the titer of the baseline sample.
Time Frame: Baseline to Week 24
Population: Immunogenicity-analysis population included all participants randomly assigned to study treatment who received any study treatment with at least one post-dose anti-drug antibody (ADA) assessment. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Satralizumab
Number analyzed (Participants) | 94
Participants
  Participants with ADA postive sample | 23
  Participants with ADA negative sample | 71

29. Secondary Outcome: Serum Concentrations of Satralizumab
Time Frame: Weeks 0, 2, 4, 8, 12, 16, 20 and 24
Population: Pharmacokinetic (PK)-evaluable population included all participants randomly assigned to study treatment who received at least one dose and had sufficient sampling to permit PK evaluation. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Satralizumab 180 mg: Participants received satralizumab 180 mg, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
Arm/Group | Satralizumab 120 mg | Satralizumab 180 mg
Number analyzed (Participants) | 87 | 9
mg
  Week 0: number analyzed (Participants) | 87 | 8
  Week 0 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not evaluable as samples were below limit of quantification. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not evaluable as samples were below limit of quantification.
  Week 2: number analyzed (Participants) | 85 | 8
  Week 2 | 9740 (5270) | 9620 (5210)
  Week 4: number analyzed (Participants) | 86 | 9
  Week 4 | 19000 (8530) | 18900 (7290)
  Week 8 | 17300 (9550) | 21700 (9690)
  Week 12: number analyzed (Participants) | 84 | 9
  Week 12 | 15600 (9030) | 19300 (13000)
  Week 16: number analyzed (Participants) | 82 | 9
  Week 16 | 15800 (9710) | 14500 (10100)
  Week 20: number analyzed (Participants) | 82 | 9
  Week 20 | 14900 (9180) | 15100 (10100)
  Week 24: number analyzed (Participants) | 83 | 9
  Week 24 | 14800 (10100) | 14800 (10900)

ADVERSE EVENTS:
Time Frame: DB Period Arms: Day 1 up to approximately 24 weeks; Overall Satralizumab Treatment (OST) Period: Participants receiving Satralizumab in DB: Day 1 in DB up to end of OLE (approximately 116 weeks); Participants receiving Placebo in DB: Day 1 in OLE up to end of OLE (approximately 92 weeks) As placebo has no active drug, all AEs for placebo (matched to 120 mg and 180 mg satralizumab) are reported together.
Description: DB Period: SE Population used;
  All Treated Participants Set=all participants who received at least 1 dose of satralizumab in DB & OLE period.
  As pre-specified in SAP, AEs were reported for DB period & OST period. OST includes data for all participants from 1st dose of satralizumab (in DB for participants receiving satralizumab & in OLE for participants receiving placebo in DB) up to 4 weeks after the last dose (if discontinued), or last contact with participant, whatever occurred first.
Groups:
- DB Period: Placebo: Participants received satralizumab matched placebo, SC, at Weeks 0, 2, 4, and Q4W thereafter until the end of the DB period.
- DB Period: Satralizumab 120mg: Participants received satralizumab 120 mg, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
- DB Period: Satralizumab 180mg: Participants received satralizumab 180 mg, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period.
- Overall Satralizumab 120mg: Participants who received satralizumab 120 mg, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period continued receiving satralizumab 120 mg, Q4W in the OLE period. Participants who received placebo in the DB period received satralizumab, 120 mg at Weeks 0, 2, and 4 (loading doses), and Q4W thereafter (maintenance doses) in the OLE period. Participants continuing satralizumab treatment from the DB period received a placebo injection on Week 2 of OLE to maintain blinding to DB treatment assignment.
- Overall Satralizumab 180mg: Participants who received satralizumab 180 mg, SC, at Weeks 0, 2, 4 (loading doses), and Q4W (maintenance doses) thereafter until the end of the DB period continued receiving satralizumab 180 mg, Q4W in the OLE period. Participants who received placebo in the DB period received satralizumab, 180 mg at Weeks 0, 2, and 4 (loading doses), and Q4W thereafter (maintenance doses) in the OLE period. Participants continuing satralizumab treatment from the DB period received a placebo injection on Week 2 of OLE to maintain blinding to DB treatment assignment.
Arm/Group | DB Period: Placebo | DB Period: Satralizumab 120mg | DB Period: Satralizumab 180mg | Overall Satralizumab 120mg | Overall Satralizumab 180mg
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/87 | 0/9 | 1/159 | 0/25
Serious Adverse Events (participants affected / at risk) | 6/92 | 3/87 | 0/9 | 18/159 | 5/25
Other Adverse Events (participants affected / at risk) | 40/92 | 48/87 | 8/9 | 95/159 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=92) | DB Period: Satralizumab 120mg (N=87) | DB Period: Satralizumab 180mg (N=9) | Overall Satralizumab 120mg (N=159) | Overall Satralizumab 180mg (N=25)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis crisis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=92) | DB Period: Satralizumab 120mg (N=87) | DB Period: Satralizumab 180mg (N=9) | Overall Satralizumab 120mg (N=159) | Overall Satralizumab 180mg (N=25)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 3 (3) | 1 (1) | 11 (11) | 1 (2)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 8 (9) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 7 (7) | 11 (11) | 1 (1) | 22 (24) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (6) | 0 (0) | 18 (23) | 2 (4)
Pharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 0 (0) | 8 (12) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 6 (7) | 0 (0) | 23 (34) | 3 (5)
Urinary tract infection (Infections and infestations) | 6 (6) | 4 (5) | 1 (1) | 13 (19) | 1 (1)
Intercepted medication error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (2) | 1 (1) | 10 (13) | 3 (4)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Weight increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 8 (8) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (4) | 2 (2) | 6 (7) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 9 (9) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 0 (0) | 6 (7) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 9 (17) | 9 (16) | 0 (0) | 20 (40) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (4) | 3 (3) | 0 (0) | 8 (8) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 2 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 8 (8) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 4 (4) | 1 (1) | 9 (10) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT04963270/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT04963270/SAP_001.pdf